CLINICAL TRIAL: NCT05311098
Title: Cryoablation With Vestibular Expansion for the Treatment of Paroxysmal/Short-course Persistent Atrial Fibrillation
Acronym: AF-PACC-CRYO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Director, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AF-PACC-CRYO
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Vestibule Group (Experimental): Cryoablation
  Interventions: Device: cryoablation

INTERVENTIONS:
Device: cryoablation — Treatment of atrial fibrillation with cryoablation catheters

SUMMARY:
The purpose of this study was to verify the safety and efficacy of routine and extended vestibular ablation in the treatment of paroxysmal/short-course persistent atrial fibrillation.

DETAILED DESCRIPTION:
The purpose of this study was to verify the safety and efficacy of routine and extended vestibular ablation using the Medtronic Arctic Front AdvanceTM catheter in the treatment of paroxysmal/short-course persistent atrial fibrillation

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ age ≤ 85 years old;
2. Patients with paroxysmal/short-term persistent atrial fibrillation;
3. Be able to understand the purpose of the research, voluntarily participate in the research and sign the informed consent.

Exclusion Criteria:

1. Echocardiography shows that the left atrium diameter is greater than or equal to 45mm;
2. Preoperative CT or esophageal echocardiography suggests that there is a thrombus in the left atrium/left atrial appendage;
3. Those who have undergone left atrial ablation or left atrial surgery;
4. Those who have received simple left atrial appendage occlusion;
5. New York heart function class (NYHA) class III or IV congestive heart failure or LVEF (%) less than 40%;
6. Those who have undergone valve repair;
7. Preoperative electrocardiogram or Holter confirmed the presence of typical atrial flutter or other supraventricular tachycardia (holding The duration is greater than 30 s);
8. Secondary atrial fibrillation, including uncontrolled hyperthyroidism, acute alcoholism, cardiac surgery postoperative atrial fibrillation, etc.;
9. History of acute coronary events or percutaneous coronary stent intervention within 6 months before enrollment;
10. Those with a history of cardioverter-defibrillator (ICD) implantation or a history of cardiac resynchronization therapy (CRT);
11. History of stroke or transient ischemic attack within 6 months before enrollment;
12. Those with obvious bleeding tendency who cannot receive postoperative systemic anticoagulation;
13. Severe structural heart disease, including moderate to severe mitral insufficiency or stenosis, previous myocardial infarction, hypertrophic cardiomyopathy, etc.;
14. Combined with other serious diseases, the life expectancy is less than 12 months;
15. Women who are pregnant, breastfeeding and planning to become pregnant;
16. Have participated in or are participating in clinical investigators of other drugs or devices within 3 months before enrollment;
17. Other conditions assessed by the investigator to be unsuitable for inclusion in this study, such as persons with mental disorders or mental disorders.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
1-year atrial fibrillation-free rate | 1-year
  Treatment success rate within 12 months after surgery (ie: no antiarrhythmic drug use, and no atrial fibrillation lasting ≥30s after a 3-month postoperative blank period to a 12-month postoperative follow-up). , AF), Atrial Flutter (AFL) or Atrial Tachycardia (AT) events).
pulmonary vein isolation rate | Immediate
  Immediate success rate of surgery: the percentage of subjects whose pulmonary veins were successfully electrically isolated at the end of surgery (including 30-minute observation time) to the total number of patients undergoing surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No